CLINICAL TRIAL: NCT03779191
Title: Phase II, Open Label, Single Arm Trial of Alectinib in Combination With Bevacizumab in Untreated and Previously Treated Patients With Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer (NSCLC) With Positive ALK Driver Mutation
Brief Title: Alectinib in Combination With Bevacizumab in ALK Positive NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Coordinator of the Thoracic Oncology Unit and Laboratory of Personalized Medicine, Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alectinib plus Bevacizumab
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: ALK Gene Rearrangement Positive; Non-Squamous Non-Small Cell Neoplasm of Lung
MeSH Terms: interventions — alectinib; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Phase II, single arm trial assessing Alectinib in combination with Bevacizumab in untreated and previously treated patients with Advanced or Metastatic Non-Squamous ALK-rearranged NSCLC
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention (Experimental): Patients in this intervention arm will receive the therapeutic combination of Alectinib dosed PO 600 mg bis in die (BID) with meals and Bevacizumab 15 mg/kg intravenously every 3 weeks until disease progression, unacceptable toxicity, or other reasons specified in the protocol
  Interventions: Drug: Alectinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Alectinib — Alectinib dosed 600 mg twice a day (BID) with meals until disease progression, unacceptable toxicity, or other reasons specified in the protocol
  Other Names: Alecensa
Drug: Bevacizumab — Bevacizumab 15 mg/kg intravenously every 3 weeks until disease progression, unacceptable toxicity, or other reasons specified in the protocol
  Other Names: Avastin

SUMMARY:
This single-arm, open-label, phase II clinical study aims to evaluate the progression-Free Survival (PFS) of the combination of Alectinib plus Bevacizumab in untreated and first and second-line chemotherapy failed subjects with stage IIIB/IV or recurrent disease after receiving radiation therapy or surgical resection.

The main question to be answered is:

Whether the combination of Alectinib plus Bevacizumab will improve PFS in untreated and previously treated subjects with advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) and positive ALK translocation.

Participants will be treated with Alectinib and Bevacizumab every three weeks until disease progression, unacceptable toxicity, or patient withdrawal of consent.

DETAILED DESCRIPTION:
Dose selection The required dose amount for Alectinib is based on a fixed dose of 600 mg, and the dose for Bevacizumab when preparing the solution is based on the subject's weight in kilograms (kg).

Dose Modification The administration of Alectinib/Bevacizumab will be stopped in case of Grade 4 hematological toxicities or Grade 3 non-hematological drug-related toxicities, including severe or life-threatening abnormalities.

The test treatment should be discontinued if toxicity does not resolve to grade 0-1 within 12 weeks after the last application.

With an adverse laboratory event still graded two, after 12 weeks, they can continue treatment at trial only if the reaction is asymptomatic and controlled.

Subjects who experience a recurrence of the same severe or life-threatening event to the same or greater degree with a re-challenge of alectinib/bevacizumab should discontinue the trial treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, ≥18 years of age.
2. Subjects with NSCLC with known ALK-rearrangement tested with FDA-approved test (IHQ or FISH).
3. Subjects with sufficient tissue to test for ALK-rearranged using IHQ or FISH.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
5. Karnofsky Performance Status of ≥70
6. Subjects with histologically confirmed Stage 3B (IIIB), 4 (IV) or recurrent NSCLC (per the 8th International Association for the Study of Lung Cancer classification, non-squamous histology, with prior systemic chemotherapy (platinum-based) given as primary therapy for advanced disease. Prior adjuvant or neoadjuvant chemotherapy is permitted as long as the last administration of the prior regimen occurred at least 3 weeks prior to enrollment. Prior treatment with ALK inhibitors is permitted as long as the last administration occurred 3 weeks prior to enrollment.
7. Subjects with CNS metastases are only eligible if the CNS metastases are adequately treated with radiotherapy and/or surgery and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 1 week prior to randomization.

   1. Patients receiving radiotherapy or radiosurgery with a dose exceeding 30 Gy will have 3 weeks for neurological stabilization before randomization.
   2. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
8. Measurable disease by CT as per RECIST 1.1 criteria.

   a. The target lesions may be located on a previously irradiated field exists if documented progression of disease (radiographic) in that site.
9. At least 12 weeks of life expectancy.
10. Signed written informed consent

    1. Patients should have a signed and dated form of written informed consent approved by the institutional committee in accordance with regulatory and institutional guidelines. This must be obtained before performing any procedure related to the protocol that are not part of the normal care of the patient.
    2. Patients must be willing and able to comply with scheduled visits, treatment program, laboratory testing including filling of questionnaires the results reported by the patient and other study requirements.
11. Reproductive Status

    1. Women with reproductive potential (WOCBP) should use contraceptive methods based on tables found in Appendix 2. When a teratogenic drug test is used, and / or a drug for which there is not enough information to assess teratogenicity (have not been conducted preclinical studies) are required to use a highly effective method of contraception (failure rate less than 1 % per year). Individual methods of contraception should be determined in consultation with the researcher.
    2. The WOCBP must have a negative pregnancy test in serum or urine (minimum sensitivity 25 IU / L or equivalent units of HCG) 24 hours before starting the investigational product.
    3. Women should not be breastfeeding.
    4. Sexually active men WOCBP should use any method of contraception with a failure rate of less than 1% per year. The investigator should review contraceptive methods and the time period during which contraception to use. Men who are sexually active with WOCBP, follow the instructions of birth control for a period of 90 days, plus the time required for the investigational drug is subject to five half-lives

Exclusion Criteria:

1. Subjects with known EGFR mutations which are sensitive to available targeted inhibitor therapy (including, but not limited to, deletions in exon 19 and exon 21 [L858R] substitution mutations) are excluded. All subjects with non-squamous histology must have been tested locally for EGFR mutation status; use of an FDA-approved test is strongly encouraged (EGFR mutation testing may be performed during the Screening Period, Non-squamous subjects with unknown or indeterminate EGFR status may not be included).
2. Subjects with untreated CNS metastases are excluded.
3. Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry and no additional therapy is required or anticipated to be required during the study period.
4. Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as Vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Treatment with other investigational drugs or other anti-cancer therapy, or treatment in another clinical trial within the past 4 weeks before start of therapy or concomitantly with this trial
6. Radiographical evidence of cavitated or necrotic tumors
7. Centrally located tumors with radiographical evidence (CT or MRI) of local invasion of major blood vessels
8. History of clinically significant hemoptysis within the past 3 months
9. History of major thrombotic or clinically relevant major bleeding event in the past 6 months.
10. Known inherited predisposition to bleeding or thrombosis
11. Medical History and Concurrent Diseases

    1. Any medical condition or serious uncontrolled or active infection with hepatitis or HIV that could be reactivated.
    2. Other concurrent malignancies requiring intervention.
    3. All toxicities attributed to a previous treatment for cancer other than alopecia or fatigue, must have resolved to Grade 1 (NCI CTCAE version 4) or baseline, prior to administration of study drug.
    4. Prior treatment with tumor vaccines or other anti-tumor immune stimulating agents.
    5. Prior treatment with Alectinib.
    6. Prior treatment with Bevacizumab
    7. Subjects with a history of interstitial lung disease.
    8. Subjects must be recovered from the effects of major surgery, traumatic injury or substantially at least 7 days before the first dose of study treatment.
12. Physical Findings and Laboratory Tests

    1. Positive for the surface antigen of hepatitis B virus (HBV HBsAg) or hepatitis C ribonucleic acid (HCV RNA) Evidence indicating acute or chronic infection
    2. Known history of positive test for Human Immunodeficiency Virus (HIV) or Acquired Immune Deficiency Syndrome (AIDS).
13. Allergies and Adverse Drug Reactions to

    1. History of severe hypersensitivity to other monoclonal antibodies.
    2. Previous history of severe hypersensitivity reaction to paclitaxel.
    3. History of allergy or intolerance (unacceptable adverse event) to components of the study drug, or herbal teas that contain Polysorbate 80.
14. Sexual and Reproductive Status

    1. WOCBP pregnant or who are nursing
    2. Women with a positive pregnancy test in recruitment or prior to administration of the study drug.
15. Other Exclusion Criteria

    1. Any other serious medical condition or uncontrolled active infection, findings on physical examination, laboratory findings, altered mental status, or psychiatric condition that, in the investigator's opinion, would limit the ability of an individual to meet the requirements of study, significantly increase the risk to the subject, or which affects the interpretability of the study results.
    2. Prisoners or subjects who are involuntarily incarcerated.
    3. Subjects who are compulsorily admitted for treatment of a mental or physical illness (eg, infectious disease). Eligibility criteria for this study were carefully considered to ensure the safety of study subjects, and to ensure that the results of the study can be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Through study completion, an average of 18 months
  PFS based on response criteria according to RECIST 1.1 in untreated and previously treated patients with Advanced or metastatic ALK-rearranged Non-Squamous NSCLC who receive treatment with Alectinib plus Bevacizumab

SECONDARY OUTCOMES:
Objective response rate | 8 weeks
  To assess the ORR, based on response criteria according to RECIST 1.1, in untreated and previously treated patients with Advanced or Metastatic ALK-rearranged Non-Squamous NSCLC who receive treatment with Alectinib plus Bevacizumab.
Brain- ORR | 8 weeks
  To assess the brain ORR, based on response criteria according RECIST 1.1, in untreated and previously treated patients with Advanced or metastatic Non-Squamous NSCLC who receive treatment with Alectinib plus Bevacizumab.
Overall survival | Through study completion, an average of 18 months
  To assess the OS in untreated and previously treated patients with Advanced or metastatic Non-Squamous ALK-rearranged NSCLC who receive treatment with Alectinib plus Bevacizumab.
Time to developing brain metastases | Through study completion, an average of 18 months
  To assess the time since inclusion until developing brain metastases in untreated and previously treated patients with Advanced or metastatic Non-Squamous ALK-rearranged NSCLC who receive treatment with Alectinib plus Bevacizumab.
Change From Baseline in Global Quality of Life (QOL), Functional Scales and Symptoms Scales as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC-QLQ-C30) During Overall Treatment | From Baseline up to Cycle 20 (each cycle is 3 weeks) Day 1.
  The EORTC QLQ C30 consists of 30 questions and includes 5 functional scales (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale; 3 symptom scales (fatigue, pain, nausea, and vomiting); and 6 single items that assess additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and financial impact. All scales and single-item measures range in scores from 0 to 100. Higher scores on the functional scales represent higher levels of functioning. Higher scores on the global health status/quality of life scale represent higher health status/quality of life. Higher scores on symptom scales/items represent a greater presence of symptoms.
Change From Baseline in Lung Cancer Symptoms as Assessed by the EORTC Quality of Life Questionnaire-Lung Cancer 13 (QLQ- LC13) During Overall Treatment | From Baseline up to Cycle 20 (each cycle is 3 weeks) Day 1.
  The EORTC QLQ LC13 consists of 13 questions and includes 1 multi-item scale and 9 single items assessing symptoms (dyspnea, cough, haemoptysis, and site-specific pain), side effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and pain medication use. The scale scores rang from 0 to 100, with higher scores indicating higher ("worse") level of symptoms.
Time to Deterioration (TTD) in Participant Reported Global Quality of Life, or Cough From QLQ-LC13 | From Baseline up to Cycle 20 (each cycle is 3 weeks) Day 1.
  The EORTC QLQ C30 consists of 30 questions and includes 5 functional scales (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale; Higher scores on the global health status/quality of life scale represent higher health status/quality of life. TTD in pain in global Quality of Life was defined as the time from randomization to the first time the participant's score showed a 10 point or greater increase after baseline in any of the 3 symptoms. TTD in months was calculated as (date of deterioration or censoring - randomization date +1)/30.4375.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar G Arrieta Rodriguez, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerología de México
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrieta O, Guzman-de Alba E, Alba-Lopez LF, Acosta-Espinoza A, Alatorre-Alexander J, Alexander-Meza JF, Allende-Perez SR, Alvarado-Aguilar S, Araujo-Navarrete ME, Argote-Greene LM, Aquino-Mendoza CA, Astorga-Ramos AM, Austudillo-de la Vega H, Aviles-Salas A, Barajas-Figueroa LJ, Barroso-Quiroga N, Blake-Cerda M, Cabrera-Galeana PA, Calderillo-Ruiz G, Campos-Parra AD, Cano-Valdez AM, Capdeville-Garcia D, Castillo-Ortega G, Casillas-Suarez C, Castillo-Gonzalez P, Corona-Cruz JF, Correa-Acevedo ME, Cortez-Ramirez SS, de la Cruz-Vargas JA, de la Garza-Salazar JG, de la Mata-Moya MD, Dominguez-Flores ME, Dominguez-Malagon HR, Dominguez-Parra LM, Dominguez-Peregrina A, Duran-Alcocer J, Enriquez-Aceves MI, Elizondo-Rios A, Escobedo-Sanchez MD, de Villafranca PE, Flores-Cantisani A, Flores-Gutierrez JP, Franco-Marina F, Franco-Gonzalez EE, Franco-Topete RA, Fuentes-de la Pena H, Galicia-Amor S, Gallardo-Rincon D, Gamboa-Dominguez A, Garcia-Andreu J, Garcia-Cuellar CM, Garcia-Sancho-Figueroa MC, Garcia-Torrentera R, Gerson-Cwilich R, Gomez-Gonzalez A, Green-Schneeweiss L, Guillen-Nunez Mdel R, Gutierrez-Velazquez H, Ibarra-Perez C, Jimenez-Fuentes E, Juarez-Sanchez P, Juarez-Ramiro A, Kelly-Garcia J, Kuri-Exsome R, Lazaro-Leon JM, Leon-Rodriguez E, Llanos-Osuna S, Llanos-Osuna S, Loyola-Garcia U, Lopez-Gonzalez JS, Lopez y de Antunano FJ, Loustaunau-Andrade MA, Macedo-Perez EO, Machado-Villarroel L, Magallanes-Maciel M, Martinez-Barrera L, Martinez-Cedillo J, Martinez-Martinez G, Medina-Esparza A, Meneses-Garcia A, Mohar-Betancourt A, Morales Blanhir J, Morales-Gomez J, Motola-Kuba D, Najera-Cruz MP, Nunez-Valencia Cdel C, Ocampo-Ocampo MA, Ochoa-Vazquez MD, Olivares-Torres CA, Palomar-Lever A, Patino-Zarco M, Perez-Padilla R, Pena-Alonso YR, Perez-Romo AR, Aquilino Perez M, Pinaya-Ruiz PM, Pointevin-Chacon MA, Poot-Braga JJ, Posadas-Valay R, Ramirez-Marquez M, Reyes-Martinez I, Robledo-Pascual J, Rodriguez-Cid J, Rojas-Marin CE, Romero-Bielma E, Rubio-Gutierrez JE, Saenz-Frias JA, Salazar-Lezama MA, Sanchez-Lara K, Sansores Martinez R, Santillan-Doherty P, Alejandro-Silva J, Tellez-Becerra JL, Toledo-Buenrostro V, Torre-Bouscoulet L, Torecillas-Torres L, Torres M, Tovar-Guzman V, Turcott-Chaparro JG, Vazquez-Cortes JJ, Vazquez-Manriquez ME, Vilches-Cisneros N, Villegas-Elizondo JF, Zamboni MM, Zamora-Moreno J, Zinser-Sierra JW. [National consensus of diagnosis and treatment of non-small cell lung cancer]. Rev Invest Clin. 2013 Mar;65 Suppl 1:S5-84. Spanish. PMID 24459776
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Spiro SG, Silvestri GA. One hundred years of lung cancer. Am J Respir Crit Care Med. 2005 Sep 1;172(5):523-9. doi: 10.1164/rccm.200504-531OE. Epub 2005 Jun 16. PMID 15961694
- [Background] Choi YL, Soda M, Yamashita Y, Ueno T, Takashima J, Nakajima T, Yatabe Y, Takeuchi K, Hamada T, Haruta H, Ishikawa Y, Kimura H, Mitsudomi T, Tanio Y, Mano H; ALK Lung Cancer Study Group. EML4-ALK mutations in lung cancer that confer resistance to ALK inhibitors. N Engl J Med. 2010 Oct 28;363(18):1734-9. doi: 10.1056/NEJMoa1007478. PMID 20979473
- [Background] Ou SH, Bartlett CH, Mino-Kenudson M, Cui J, Iafrate AJ. Crizotinib for the treatment of ALK-rearranged non-small cell lung cancer: a success story to usher in the second decade of molecular targeted therapy in oncology. Oncologist. 2012;17(11):1351-75. doi: 10.1634/theoncologist.2012-0311. Epub 2012 Sep 18. PMID 22989574
- [Background] Soda M, Choi YL, Enomoto M, Takada S, Yamashita Y, Ishikawa S, Fujiwara S, Watanabe H, Kurashina K, Hatanaka H, Bando M, Ohno S, Ishikawa Y, Aburatani H, Niki T, Sohara Y, Sugiyama Y, Mano H. Identification of the transforming EML4-ALK fusion gene in non-small-cell lung cancer. Nature. 2007 Aug 2;448(7153):561-6. doi: 10.1038/nature05945. Epub 2007 Jul 11. PMID 17625570
- [Background] Inamura K, Takeuchi K, Togashi Y, Nomura K, Ninomiya H, Okui M, Satoh Y, Okumura S, Nakagawa K, Soda M, Choi YL, Niki T, Mano H, Ishikawa Y. EML4-ALK fusion is linked to histological characteristics in a subset of lung cancers. J Thorac Oncol. 2008 Jan;3(1):13-7. doi: 10.1097/JTO.0b013e31815e8b60. PMID 18166835
- [Background] Doebele RC, Pilling AB, Aisner DL, Kutateladze TG, Le AT, Weickhardt AJ, Kondo KL, Linderman DJ, Heasley LE, Franklin WA, Varella-Garcia M, Camidge DR. Mechanisms of resistance to crizotinib in patients with ALK gene rearranged non-small cell lung cancer. Clin Cancer Res. 2012 Mar 1;18(5):1472-82. doi: 10.1158/1078-0432.CCR-11-2906. Epub 2012 Jan 10. PMID 22235099
- [Background] Pulford K, Lamant L, Morris SW, Butler LH, Wood KM, Stroud D, Delsol G, Mason DY. Detection of anaplastic lymphoma kinase (ALK) and nucleolar protein nucleophosmin (NPM)-ALK proteins in normal and neoplastic cells with the monoclonal antibody ALK1. Blood. 1997 Feb 15;89(4):1394-404. PMID 9028963